CLINICAL TRIAL: NCT03206710
Title: Maternal Vitamin C Supplementation to Decrease Effects of Smoking During Pregnancy on Infant Lung Function and Health: Follow-up of 2 Randomized Trials and Association With Changes in DNA Methylation
Brief Title: Vitamin C Supplementation to Pregnant Smokers: Follow-up of 2 Randomized Trials Plus Changes in DNA Methylation
Acronym: VCSIP-ECHO
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Indiana University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Cynthia McEvoy, MD, MCR, Oregon Health and Science University
Other Study IDs: VCSIP ECHO; UG3OD023288 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Asthma; Wheezing; In Utero Nicotine; Pulmonary Function
Keywords: vitamin C; ascorbic acid; wheeze; nicotine; smoke exposure; long term follow up; pulmonary function testing; forced expiratory flows
MeSH Terms: conditions — Asthma; Respiratory Sounds

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buccal swabs, hair, blood, and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- smokers who received Vitamin C
  Interventions: Other: No current intervention
- smokers who received placebo
  Interventions: Other: No current intervention
- control group non-smokers
  Interventions: Other: No current intervention

INTERVENTIONS:
Other: No current intervention — This is a follow-up of two randomized trials. No active intervention is being given in the follow-up

SUMMARY:
In a randomized clinical trial (RCT) published in JAMA, the investigators have provided evidence that vitamin C supplementation (500 mg daily during pregnancy) ameliorates the effects of maternal smoking during pregnancy on offspring lung function and subsequent incidence of wheeze by 48% through 1 year of age. The investigators are currently completing a second RCT of vitamin C supplementation in pregnant smokers with more robust measures of pulmonary outcomes. The purpose of this ECHO application is to combine these 2 focused, interventional cohorts to allow critical longitudinal follow-up of respiratory outcomes in these children including the study of pulmonary function test (PFT) trajectories and incidence of recurrent wheeze/asthma from infancy through early adolescence in offspring of pregnant smokers randomized to vitamin C versus placebo.

DETAILED DESCRIPTION:
In a randomized clinical trial (RCT) published in JAMA, the investigators have provided evidence that vitamin C supplementation (500 mg daily during pregnancy) ameliorates the effects of maternal smoking during pregnancy on offspring lung function and subsequent incidence of wheeze by 48% through 1 year of age. the investigators are currently completing a second RCT of vitamin C supplementation in pregnant smokers with more robust measures of pulmonary outcomes. The purpose of this ECHO application is to combine these 2 focused, interventional cohorts to allow critical longitudinal follow-up of respiratory outcomes in these children including the study of pulmonary function test (PFT) trajectories and incidence of recurrent wheeze/asthma from infancy through early adolescence in offspring of pregnant smokers randomized to vitamin C versus placebo.

This will allow the investigators to study the duration of the protection vitamin C provides in the face of in-utero smoke, the relationship between PFTs and the development of recurrent wheeze and/or asthma. In addition we have preliminary data suggesting that, in parallel with the effects of vitamin C on the reduction of pulmonary harm, the supplementary vitamin C blocked the majority of significant changes in DNA methylation induced by maternal smoking in placentas, cord blood and offspring cheek cells. Thus this study will also study the association between the prevention of wheeze/asthma associated with maternal smoking during pregnancy and the prevention of epigenetic changes caused by maternal smoking during pregnancy. By linking the clinical outcomes of decreased wheeze/asthma and pulmonary function in offspring of smokers to epigenetic changes, this study has the potential to identify genes linked to the effects of maternal smoking on lung development and the protective effects of vitamin C.

ELIGIBILITY:
Inclusion Criteria:

* Women and their offspring randomized to vitamin C versus placebo during pregnancy in VCSIP1 or VCSIP2 as well as pregnant nonsmokers and their offspring enrolled as the reference group in VCSIP 1 or VCSIP2

Exclusion Criteria:

* Patients specifically withdrawing consent from VCSIP1 or VCSIP2

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study is a follow-up of women and their offspring who previously participated in NCT00632476 and/or NCT01723696.
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Improved pulmonary function | through 15 years of age
  The first primary aim of this study is to demonstrate improved pulmonary function trajectories as measured with forced expiratory flows through 15 years of age in the offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo.
Decreased recurrent wheeze/asthma | through 15 years of age
  The second primary aim of this study is to demonstrate a decreased incidence of recurrent wheeze/ asthma through 15 years of age in the offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo.

SECONDARY OUTCOMES:
Decreased incidence of recurrent wheeze/asthma | through 15 years of age
  A secondary aim of this study is to demonstrate a decreased incidence of recurrent wheeze/asthma through 15 years of age in offspring of pregnant smokers randomized to vitamin C (500 mg/day) versus placebo
Epigenetic changes | through 15 years of age
  An additional secondary aim of the study is the analysis of epigenetic changes caused by maternal smoking and reversed by vitamin C at birth. DNA methylation will be measured in biologic samples and then followed longitudinally through ages 15.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Oregon Health and Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McEvoy CT, Schilling D, Clay N, Jackson K, Go MD, Spitale P, Bunten C, Leiva M, Gonzales D, Hollister-Smith J, Durand M, Frei B, Buist AS, Peters D, Morris CD, Spindel ER. Vitamin C supplementation for pregnant smoking women and pulmonary function in their newborn infants: a randomized clinical trial. JAMA. 2014 May;311(20):2074-82. doi: 10.1001/jama.2014.5217. PMID 24838476